CLINICAL TRIAL: NCT06457971
Title: Clinical Assessment Protocol: Anovo Surgical System in Ventral Hernia
Brief Title: Anovo Surgical System in Ventral Hernia
Acronym: CLEVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Momentis Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEMIC-12219
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic Ventral Hernia (Experimental): Subjects undergoing robotic ventral hernia with the Anovo Surgical System.
  Interventions: Device: Robotic Ventral Hernia Repair

INTERVENTIONS:
Device: Robotic Ventral Hernia Repair — The AnovoTM Surgical System is an endoscopic instrument control system that is intended to assist in the accurate control of the Instrument ARMS with graspers and electrosurgery devices for endoscopic manipulation of tissue including grasping, blunt dissection, approximation, and electrosurgery, during single site, laparoscopic surgical procedures. The AnovoTM System's articulated robotic arms allow the surgeon to access and reach different structures in the pelvic and abdominal cavity. Closing the fascial defect robotically is easier from a technical standpoint than attempting it with classical laparoscopic instruments

SUMMARY:
The study is aimed to clinically assess the AnovoTM Surgical System in ventral hernia procedures. Extensive preclinical testing of the system's integrity and safety has been performed to assure adequate safety for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old.
* Subjects able to provide written informed consent.
* Subject deemed eligible candidate by surgeon and will comply with the study procedures.
* Subjects with ventral hernia.
* Subjects with ASA grade I to III.
* Subject must sign and date informed consent prior to treatment.
* Subject can undergo general anesthesia per anesthesiologist assessment.

Exclusion Criteria:

* Women who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical investigation.
* Subject has medical condition, which in the judgement of the investigator makes the subject a poor candidate for the investigational procedure.
* Participation in another clinical trial that is in the active phase.
* Subject unwilling or inability to follow procedures outlined in the protocol.
* Subjects who are not suitable for robotic surgery, the Subject will be excluded from the study and the will be considered a screen failure and the surgeon will proceed with a standard multiport laparoscopic Hernia repair.
* Subjects who present any adverse event before use the Anovo Surgical System ("Anovo") that can affect evaluation of safety and performance of Investigational Device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Conversion | Intra-Operative
  The primary endpoint is rate of conversion to open surgery or multiport laparoscopic approach. As this is a clinical assessment, no pre-determined success criteria have been set.

SECONDARY OUTCOMES:
IntraOperative Procedural Outcomes - AE and SADE | Intra-Operative
  IntraOperative Adverse and Serious Adverse Events
IntraOperative Procedural Outcomes - Device/Procedure AE | Intra-Operative
  IntraOperative device related and / or procedure related Adverse Event
IntraOperative Procedural Outcomes - Time | Intra-Operative
  IntraOperative Operative Time
Post Operative Procedural Outcomes - AE and SADE | Through study completion, an average of 4 weeks.
  Post operative procedural outcomes such as Adverse and Serious Adverse Events and Series Adverse Device Effects
Post Operative Procedural Outcomes - Wound Seroma | Through study completion, an average of 4 weeks.
  Post operative procedural outcomes such as post operative wound seroma
Post Operative Procedural Outcomes - SSI | Through study completion, an average of 4 weeks.
  Post operative procedural outcomes such as surgical site infection
Post Operative Procedural Outcomes - Length of Stay | Through hospital discharge, up to approximately 3 days
  Post operative procedural outcomes such as length of hospital stay
Procedure Completion | Intra-Operative
  Rate of procedure completion with the device
Console Time | Intra-Operative
  Length of time the surgeon is actively using the surgeon console to control the robotic device
Docking Time | Intra-Operative
  Length of time spent docking the robotic device, described as when the robotic instrument arms are inserted through the cannula.
Draping Time | Intra-Operative
  Length of time spent draping the robotic device

CONTACTS AND LOCATIONS:
Locations (2):
- Imelda Hospital, Bonheiden, Belgium
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No